CLINICAL TRIAL: NCT06575699
Title: Rectus Sheath Block With Liposomal Bupivacaine for Postoperative Analgesia Following Gynecologic Oncology Surgery: A Pilot Study
Brief Title: Rectus Sheath Block for Analgesia After Gynecological Laparotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00115981
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Gynecologic Surgical Procedures
MeSH Terms: interventions — Tea; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rectus Sheath Block Group (Prospective arm) (Experimental): Thirty subjects will be prospectively enrolled and will receive a bilateral rectus sheath block under ultrasound guidance using 133 mg liposomal bupivacaine and 20 ml bupivacaine 0.25% per side.
  Interventions: Procedure: Rectus sheath block; Drug: Liposomal bupivacaine; Drug: Bupivacaine Hydrochloride
- Thoracic Epidural Analgesia Group (retrospective arm) (Active Comparator): 60 patients who received thoracic epidural analgesia as part of our enhanced recovery after surgery protocol and stayed in hospital for at least 72 h.
  Interventions: Procedure: Thoracic Epidural Analgesia; Drug: Bupivacaine-Hydromorphone Cassette

INTERVENTIONS:
Procedure: Rectus sheath block — bilateral rectus sheath block under ultrasound guidance using 133 mg liposomal bupivacaine and 20 ml bupivacaine 0.25% per side deposited between the rectus abdomens muscle and the posterior rectus sheath.
  Arms: Rectus Sheath Block Group (Prospective arm)
Procedure: Thoracic Epidural Analgesia — Low thoracic Epidural Analgesia.
  Arms: Thoracic Epidural Analgesia Group (retrospective arm)
Drug: Liposomal bupivacaine — 133 mg liposomal bupivacaine per side for rectus sheath block
  Arms: Rectus Sheath Block Group (Prospective arm)
Drug: Bupivacaine Hydrochloride — 20 mL bupivacaine 0.25% per side for rectus sheath block
  Arms: Rectus Sheath Block Group (Prospective arm)
Drug: Bupivacaine-Hydromorphone Cassette — Bupivacaine 0.625% with hydromorphone 10 mcg/ml for the epidural solution
  Arms: Thoracic Epidural Analgesia Group (retrospective arm)

SUMMARY:
Thirty subjects undergoing laparotomy for Gynecologic oncology surgery will be prospectively enrolled and will receive a bilateral rectus sheath block (RSB) under ultrasound guidance using 133 mg liposomal bupivacaine and 20 ml bupivacaine 0.25% per side. Cases will be matched in a 1:2 ratio by age, race, insurance status and duration of surgery with historical controls who received postoperative analgesia using thoracic epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years presenting for a laparotomy for Gynecologic malignancy with a vertical incision.
2. ASA Classification II or III.
3. English speaking patients

Exclusion Criteria:

1. BMI >50 kg/m2.
2. Chronic pain or chronic opioid therapy.
3. Allergy or contraindication to local anesthetics or any component of the multimodal analgesic regimen (NSAIDs and acetaminophen)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption 0- 72 hours after surgery | 0-72 hours after time 0 (end of surgery)

SECONDARY OUTCOMES:
Total postsurgical opioid consumption at 0-24, 24-48, and 48-72 hours | 0-24 hours, 24-48 hours and 48-72 hours after time 0 (end of surgery)
Number of patients with intraoperative hypotension | Intraoperative
Number of patients with postoperative hypotension | 0-72 hours after time 0 (end of surgery)
Number of patients receiving rescue antiemetics | 0-72 hours after time 0 (end of surgery)
Number of patients receiving rescue antipruritics | 0-72 hours after time 0 (end of surgery)
Number of patients developing ileus or constipation | 0-72 hours after time 0 (end of surgery)
Number of patients with respiratory Depression | 0-72 hours after time 0 (end of surgery)
Area under the curve (AUC) of visual analog scale (VAS) pain intensity scores through 72 hours (AUC0-72) | 0-72 hours after time 0 (end of surgery)
  Visual analog scores 0-10 (0=no pain, 10=worst possible pain)
Maximum pain scores reported | 0-72 hours after time 0 (end of surgery)
  Visual analog scores 0-10 (0=no pain, 10=worst possible pain)
Time to mobilization | 0-72 hours after time 0 (end of surgery)
Time to urinary catheter removal | 0-72 hours after time 0 (end of surgery)
Duration of post anesthesia care unit (PACU) stay | 0-6 hours after time 0 (end of surgery)
Duration of hospital stay | 0-10 days after surgery
Number of patients receiving intraoperative vasopressors | Intraoperative

OTHER OUTCOMES:
Complications related to rectus sheath block or epidural analgesia | 0-72 hours after time 0 (end of surgery)
  Inadvertent dural puncture, postdural puncture headache, need to discontinue epidural due to hypotension, epidural hematoma.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Habib, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon reasonable request